CLINICAL TRIAL: NCT06907745
Title: Splintless Virtual Surgical Plan with Mandible-first Technique in Orthognathic Surgery: Tridimensional Accuracy Analysis
Brief Title: Splintless Virtual Surgical Plan with Mandible-first Technique: 3D Accuracy Analysis
Acronym: MandiFirst
Status: Recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: Mandible First
Record Dates: First submitted 2024-05-18; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-06

CONDITIONS: Dentofacial Deformities
MeSH Terms: conditions — Dentofacial Deformities

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Bimaxillary Osteotomy — Maxillary LeFort I osteotomy and mandible osteotomy (BSSO) without intermediate splint.

SUMMARY:
Accuracy assessment through three-dimensional superposition of the post-operative volumetric CT and the digital therapeutic project files.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age over 18 and under 60
* Diagnosis of dento-skeletal dysmorphosis involving the middle third and lower part of the face
* Patients with consent to surgery
* Patients in good general health according to the evaluation of the PI and on the basis of the anamnesis and clinical examination

Exclusion Criteria:

* History of previous maxillomandibular fracture
* Treatment with anticoagulant drugs
* Treatment with intravenous bisphosphonates
* Treatment with anticonvulsants
* Patient's inability to maintain home hygiene standards in accordance with the study requirements
* History of drug and/or alcohol abuse
* Chronic corticosteroid therapy
* Radiotherapy, chemotherapy and/or immunosuppressive treatment or radiotherapy in the last 5 years
* Psychosis
* Pregnant or breastfeeding
* Poor compliance
* Endocrinological disorders in poor pharmacological control
* Other uncontrolled systemic conditions that preclude performing surgical procedures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diagnosis of dentoskeletal disorders
Sampling Method: Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy evaluation | 1 month post-op
  3D superposition of post-operative volumetric CT and the digital therapeutic project files.
  The variables and parameters analysis will be performed after the data distribution analysis, using the D'Agostino Pearson omnibus normality test: normal distribution data will be expressed as mean and standard deviation; non-normal distribution data will be expressed as median and interquartile range.
  The quantitative and qualitative variables will be expressed in terms of absolute frequencies and percentage value.
  Image superposition accuracy will be defined by measuring distances between the different anatomical reference points, considering excellent accuracy for distances less than 2 mm. Correlation and multivariate analysis models will be developed to define the secondary outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale Galeazzi-Sant'Ambrogio, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Scientific Pubblication